CLINICAL TRIAL: NCT01199705
Title: A Multicenter Study of Efficacy, Safety, Tolerability, and Pharmacokinetics of Immune Globulin Subcutaneous (Human) IgPro20 in Subjects With Primary Immunodeficiency
Brief Title: Study of Subcutaneous Immune Globulin in Patients Requiring IgG Replacement Therapy (Japan Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZLB06_002CR; U1111-1116-6379 (Other: WHO Universal Trial Number)
Record Dates: First submitted 2010-09-08; First posted 2010-09-13 (Estimated); Results first posted 2013-03-20 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2013-03

CONDITIONS: Primary Immune Deficiency
Keywords: Immune globulin subcutaneous; SCIG; Primary immunodeficiency; PID
MeSH Terms: conditions — Primary Immunodeficiency Diseases | interventions — gamma-Globulins; Hizentra

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IgPro20 (Experimental)
  Interventions: Biological: Immune Globulin Subcutaneous (Human) (SCIG)

INTERVENTIONS:
Biological: Immune Globulin Subcutaneous (Human) (SCIG) — IgPro20 is a 20% (weight per volume [w/v]) liquid formulation of human SCIG. Subjects will receive weekly infusions of IgPro20 at a weekly dosage calculated based on previous IVIG treatment.
  Other Names: Hizentra

SUMMARY:
The objective of this study is to assess the efficacy, safety, tolerability, and pharmacokinetics of a subcutaneous immune globulin (SCIG; IgPro20) in subjects with primary immunodeficiency (PID). In addition, the study will assess the health-related quality of life and pharmacoeconomic aspects related to treatment with IgPro20.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PID with hypo- or agammaglobulinemia requiring IgG replacement therapy
* Intravenous IgG (IVIG) therapy at regular 3- or 4-week intervals at a stable dose for at least 3 doses prior to signing of informed consent
* Written informed consent

Exclusion Criteria:

* Newly diagnosed PID, i.e., subjects who have not previously received immunoglobulin replacement therapy
* Ongoing serious bacterial infections (SBIs: pneumonia, bacteremia/septicemia, osteomyelitis/septic arthritis, bacterial meningitis, or visceral abscess) at the time of screening
* Ongoing or history of concomitant malignancies of lymphoid cells such as lymphocytic leukemia, non-Hodgkin's lymphoma, and immunodeficiency with thymoma
* Allergic or other severe reactions to immunoglobulins or other blood products recorded in the past 3 months or at the time of screening
* Pregnancy or nursing mother
* A positive result at screening on any of the following viral markers: human immunodeficiency virus-1 (HIV-1), HIV-2, hepatitis C virus, or hepatitis B virus
* Participation in a study with other investigational product during this study and within 3 months prior to screening
* Subjects who donated blood (200 mL within one month or 400 mL within 3 months prior to screening), or planning to donate blood during the study

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-09; Primary Completion 2011-08 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yoriyuki Shiga, Study Director — CSL Behring K.K.
Locations (10):
- Japan (10):
  - Study site, Nagoya, Aichi Pref.
  - Study site, Chiba, Chiba Pref.
  - Study site, Gifu, Gifu Pref.
  - Study site, Sapporo, Hokkaido
  - Study site, Sendai, Miyagi Pref.
  - Study site, Fukuoka City, Osaka
  - Study site, Moriguchi, Osaka
  - Study site, Osaka, Osaka
  - Study site, Koshigaya, Saitama Pref.
  - Study site, Tokorozawa, Saitama Pref.

REFERENCES:
- [Background] Igarashi A, Kanegane H, Kobayashi M, Miyawaki T, Tsutani K. Cost-minimization analysis of IgPro20, a subcutaneous immunoglobulin, in Japanese patients with primary immunodeficiency. Clin Ther. 2014 Nov 1;36(11):1616-24. doi: 10.1016/j.clinthera.2014.08.007. Epub 2014 Sep 16. PMID 25236916
- [Result] Kanegane H, Imai K, Yamada M, Takada H, Ariga T, Bexon M, Rojavin M, Hu W, Kobayashi M, Lawo JP, Nonoyama S, Hara T, Miyawaki T. Efficacy and safety of IgPro20, a subcutaneous immunoglobulin, in Japanese patients with primary immunodeficiency diseases. J Clin Immunol. 2014 Feb;34(2):204-11. doi: 10.1007/s10875-013-9985-z. Epub 2014 Feb 7. PMID 24504846

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter study enrolled subjects at nine of the participating study centers in Japan.
Pre-assignment Details: Screening took place 3 to 4 weeks prior to or at the first intravenous immunoglobulin (IVIG) infusion in the IVIG period of the study.
Groups:
- IgPro20: Immune Globulin Subcutaneous (Human): IgPro20 is a 20% (weight per volume [w/v]) liquid formulation of human immunoglobulin for subcutaneous use. Subjects will receive weekly infusions of IgPro20 at a weekly dosage calculated based on previous IVIG treatment.
Period: IVIG Treatment
Arm/Group | IgPro20
Started | 25
Completed | 25
Not Completed | 0
Period: SCIG Treatment (Wash-in/Wash-out)
Arm/Group | IgPro20
Started | 25
Completed | 24
Not Completed | 1
Not completed — Transfer of Residence | 1
Period: SCIG Treatment (Efficacy)
Arm/Group | IgPro20
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | IgPro20
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: Years] | 20.6 (13.23)
Age, Customized [Number; unit: Participants]
  < 2 years | 0
  ≥ 2 to < 12 years | 7
  ≥ 12 to ≤ 16 years | 4
  > 16 to < 65 years | 14
  ≥ 65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 16
Primary Immunodeficiency Type [Number; unit: Participants]
  Common Variable Immunodeficiency (CVID) | 10
  X-Linked Agammaglobulinemia (XLA) | 13
  Autosomal Recessive Agammaglobulinemia (ARAG) | 1
  Hyper-Immunoglobulin M (IgM) Syndrome | 1

OUTCOME MEASURES:

1. Primary Outcome: IgG Trough Level
Description: Geometric means of trough levels measured before 3 intravenous immunoglobulin (IVIG) infusions was compared with those of trough levels measured at steady-state for 3 subcutaneous immunoglobulin (SCIG) infusions (weeks 16, 20 and 24). The ratio of these geometric means was the primary outcome measure.
Time Frame: During IVIG period (IV 1, IV 2, IV 3) and during SCIG period at weeks 16, 20, and 24
Population: The PPS comprised all subjects with the disease under study who fulfilled the protocol-specified criteria for a) immunoglobulin treatment prior to and during the study, b) availability of evaluable serum IgG levels, and c) dose stability. The FAS comprised all subjects treated with IgPro20 during the efficacy period who had the disease under study.
Measure: Number (90% Confidence Interval); unit: Ratio of Geometric Means
Groups:
- IgPro20 - Per Protocol Set (PPS): The PPS data set comprised all subjects with the disease under study who fulfilled the protocol-specified criteria for a) uniformly repeated immunoglobulin treatment prior to and during the study, b) availability of evaluable serum IgG levels, and c) dose stability.
- IgPro20 - Full Analysis Set (FAS): The FAS comprised all subjects treated with IgPro20 during the SCIG efficacy period (weeks 13 to 24) who had the disease under study.
Arm/Group | IgPro20 - Per Protocol Set (PPS) | IgPro20 - Full Analysis Set (FAS)
Number analyzed (Participants) | 21 | 24
Ratio of Geometric Means | 1.09 [1.06 to 1.13] | 1.11 [1.08 to 1.15]

2. Secondary Outcome: Number of Infection Episodes (Serious and Non-serious) by Study Period
Description: Number of infection episodes (serious and non-serious) presented by study period:
  * IVIG treatment: Study subjects were treated with their IVIG therapy with 3- or 4-weekly schedules for 3 dosing cycles (9 to 12 weeks; before being switched to SCIG treatment with IgPro20).
  * SCIG treatment (wash-in/wash-out; weeks 1 to 12): IgPro20 was administered subcutaneously with the first subcutaneous (SC) IgPro20 infusion starting 1 week after the last IVIG dose. Subjects were treated with weekly SC IgPro20 infusions for a 12-week wash-in/wash-out period. The IgPro20 dose was to be equal to the weekly equivalent dose of the previous IVIG therapy.
  * SCIG treatment (efficacy; weeks 13 to 24): After the SCIG wash-in/wash-out treatment, subjects were treated with weekly SC IgPro20 infusions for a 12-week efficacy period. The IgPro20 dose was to be equal to the weekly equivalent dose of the previous IVIG therapy.
Time Frame: Up to 36 weeks
Measure: Number; unit: Number of infection episodes
Groups:
- IgPro20 - Per Protocol Set (PPS): The PPS comprised all subjects with the disease under study who fulfilled the protocol-specified criteria for a) immunoglobulin treatment prior to and during the study, b) availability of evaluable serum IgG levels, and c) dose stability.
- IgPro20 - Full Analysis Set (FAS): The FAS comprised all subjects treated with IgPro20 during the efficacy period who had the disease under study.
Arm/Group | IgPro20 - Per Protocol Set (PPS) | IgPro20 - Full Analysis Set (FAS)
Number analyzed (Participants) | 21 | 24
Number of infection episodes
  IVIG Treatment | 19 | 22
  SCIG IgPro20 Treatment (Wash-in/Wash-out) | 28 | 32
  SCIG IgPro20 Treatment (Efficacy) | 15 | 18

3. Secondary Outcome: Rate of Infection Episodes (Serious and Non-serious) by Study Period, PPS Population
Description: The annualized rate of infection episodes (serious and non-serious) was based on the total number of infection episodes and the total number of subject study days for all subjects in the specified study periods (listed below) and analysis population and adjusted to 365 days.
  Study periods:
  * IVIG treatment (up to 12 weeks)
  * SCIG IgPro20 treatment (wash-in/wash-out period) (12 weeks)
  * SCIG IgPro20 treatment (efficacy) (12 weeks)
Time Frame: Up to 36 weeks
Population: The PPS comprised all subjects with the disease under study who fulfilled the protocol-specified criteria for a) immunoglobulin treatment prior to and during the study, b) availability of evaluable serum IgG levels, and c) dose stability.
Measure: Number; unit: Infections per subject year
Units Other Than Participants: Subject Study Days
Groups:
- IVIG Treatment: Study subjects were treated with their IVIG therapy with 3- or 4-weekly schedules for 3 dosing cycles (9 to 12 weeks).
- SCIG Treatment (Wash-in/Wash-out): Weekly SC IgPro20 infusions for a 12-week wash-in/wash-out period. The IgPro20 dose was to be equal to the weekly equivalent dose of the previous IVIG therapy.
- SCIG Treatment (Efficacy): Weekly SC IgPro20 infusions for a 12-week efficacy period. The IgPro20 dose was to be equal to the weekly equivalent dose of the previous IVIG therapy.
Arm/Group | IVIG Treatment | SCIG Treatment (Wash-in/Wash-out) | SCIG Treatment (Efficacy)
Number analyzed (Participants) | 21 | 21 | 21
Number analyzed (Subject Study Days) | 1209 | 1764 | 1840
Infections per subject year | 5.74 | 5.79 | 2.98

4. Secondary Outcome: Rate of Infection Episodes (Serious and Non-serious) by Study Period, FAS Population
Description: as for outcome 3
Time Frame: Up to 36 weeks
Population: The FAS comprised all subjects treated with IgPro20 during the efficacy period who had the disease under study.
Measure: Number; unit: Infections per subject year
Units Other Than Participants: Subject Study Days
Groups:
- IVIG Treatment: Subjects were treated with their IVIG therapy with 3- or 4-weekly schedules for 3 dosing cycles (9 to 12 weeks).
Arm/Group | IVIG Treatment | SCIG Treatment (Wash-in/Wash-out) | SCIG Treatment (Efficacy)
Number analyzed (Participants) | 24 | 24 | 24
Number analyzed (Subject Study Days) | 1396 | 2016 | 2095
Infections per subject year | 5.75 | 5.79 | 3.14

5. Other Pre Specified Outcome: Annualized Rate of Serious Bacterial Infections (SBIs), PPS Population
Description: The annualized rate was based on the total number of SBIs and the total number of subject study days for all subjects in the specified study periods (listed below) and analysis population and adjusted to 365 days.
  Study periods:
  * IVIG treatment (up to 12 weeks)
  * SCIG IgPro20 treatment (wash-in/wash-out; 12 weeks)
  * SCIG IgPro20 treatment (efficacy; 12 weeks)
Time Frame: Up to 36 weeks
Population: as for outcome 3
Measure: Number; unit: SBIs per subject year
Units Other Than Participants: Subject Study Days
Groups:
- SCIG IgPro20 Treatment (Wash-in/Wash-out): Weekly SC IgPro20 infusions for a 12-week wash-in/wash-out period.
- SCIG IgPro20 Treatment (Efficacy): Weekly SC IgPro20 infusions for a 12-week efficacy period.
Arm/Group | IVIG Treatment | SCIG IgPro20 Treatment (Wash-in/Wash-out) | SCIG IgPro20 Treatment (Efficacy)
Number analyzed (Participants) | 21 | 21 | 21
Number analyzed (Subject Study Days) | 1209 | 1764 | 1840
SBIs per subject year | 0.00 | 0.00 | 0.00
Statistical Analysis 1: Comparison: IVIG Treatment; Test type: Superiority or Other; Annualized Rate = 0.00, 99% CI 1-sided [upper limit 1.390]
Statistical Analysis 2: Comparison: SCIG IgPro20 Treatment (Wash-in/Wash-out); Test type: Superiority or Other; Annualized Rate = 0.00, 99% CI 1-sided [upper limit 0.953]
Statistical Analysis 3: Comparison: SCIG IgPro20 Treatment (Efficacy); Test type: Superiority or Other; Annualized Rate = 0.00, 99% CI 1-sided [upper limit 0.914]

6. Secondary Outcome: Number of Days Out of Work/School/Kindergarten/Day Care or Unable to Perform Normal Daily Activities Due to Infections by Study Period
Description: Median number of days out of work/school/kindergarten/day care or unable to perform normal daily activities due to infections, presented by study period: IVIG treatment (up to 12 weeks), SCIG IgPro20 treatment (wash-in/wash-out; 12 weeks), and SCIG IgPro20 treatment (efficacy; 12 weeks).
Time Frame: Up to 36 weeks
Measure: Median (Full Range); unit: Days
Arm/Group | IgPro20 - Per Protocol Set (PPS) | IgPro20 - Full Analysis Set (FAS)
Number analyzed (Participants) | 21 | 24
Days
  IVIG Treatment | 0 [0 to 8] | 0 [0 to 8]
  SCIG IgPro20 Treatment (Wash-in/Wash-out) | 0 [0 to 9] | 0 [0 to 9]
  SCIG IgPro20 Treatment (Efficacy) | 0 [0 to 8] | 0 [0 to 8]

7. Other Pre Specified Outcome: Annualized Rate of Serious Bacterial Infections (SBIs), FAS Population
Description: as for outcome 5
Time Frame: Up to 36 weeks
Population: The FAS comprised all subjects treated with IgPro20 during the efficacy period who had the disease under study.
Measure: Number; unit: SBIs per subject year
Units Other Than Participants: Subject Study Days
Arm/Group | IVIG Treatment | SCIG IgPro20 Treatment (Wash-in/Wash-out) | SCIG IgPro20 Treatment (Efficacy)
Number analyzed (Participants) | 24 | 24 | 24
Number analyzed (Subject Study Days) | 1396 | 2016 | 2095
SBIs per subject year | 0.00 | 0.00 | 0.00
Statistical Analysis 1: Comparison: IVIG Treatment; Test type: Superiority or Other; Annualized Rate = 0.00, 99% CI 1-sided [upper limit 1.204]
Statistical Analysis 2: Comparison: SCIG IgPro20 Treatment (Wash-in/Wash-out); Test type: Superiority or Other; Annualized Rate = 0.00, 99% CI 1-sided [upper limit 0.834]
Statistical Analysis 3: Comparison: SCIG IgPro20 Treatment (Efficacy); Test type: Superiority or Other; Annualized Rate = 0.00, 99% CI 1-sided [upper limit 0.802]

8. Secondary Outcome: Number of Days of Hospitalization Due to Infections by Study Period
Description: Median number of days of hospitalization due to infections, presented by study period: IVIG treatment (up to 12 weeks), SCIG IgPro20 treatment (wash-in/wash-out; 12 weeks), and SCIG IgPro20 treatment (efficacy; 12 weeks).
Time Frame: Up to 36 weeks
Measure: Median (Full Range); unit: Days
Arm/Group | IgPro20 - Per Protocol Set (PPS) | IgPro20 - Full Analysis Set (FAS)
Number analyzed (Participants) | 21 | 24
Days
  IVIG Treatment | 0 [0 to 1] | 0 [0 to 1]
  SCIG IgPro20 Treatment (Wash-in/Wash-out) | 0 [0 to 0] | 0 [0 to 0]
  SCIG IgPro20 Treatment (Efficacy) | 0 [0 to 3] | 0 [0 to 3]

9. Secondary Outcome: Duration of Use of Antibiotics for Infection Prophylaxis and Treatment
Description: Median number of days of use of antibiotics for infection prophylaxis and/or treatment, presented by study period: IVIG treatment (up to 12 weeks), SCIG IgPro20 treatment (wash-in/wash-out; 12 weeks), and SCIG IgPro20 treatment (efficacy; 12 weeks).
Time Frame: Up to 36 weeks
Measure: Median (Full Range); unit: Days
Arm/Group | IgPro20 - Per Protocol Set (PPS) | IgPro20 - Full Analysis Set (FAS)
Number analyzed (Participants) | 21 | 24
Days
  IVIG Treatment | 48.5 [2 to 64] | 48.0 [2 to 64]
  SCIG IgPro20 Treatment (Wash-in/Wash-out) | 49.0 [3 to 86] | 35.5 [2 to 86]
  SCIG IgPro20 Treatment (Efficacy) | 71.0 [6 to 85] | 71.0 [6 to 85]

10. Secondary Outcome: Rate of All Adverse Events by Relatedness and Seriousness
Description: The rate of adverse events (AEs) was the number of treatment-emergent AEs over the number of infusions administered. At least possibly related AEs included possibly related AEs, probably related AEs, and related AEs.
Time Frame: For the duration of the study, up to 36 weeks
Population: The safety data set (SDS) comprised all subjects treated with the study drug.
Measure: Number; unit: AEs per infusion
Units Other Than Participants: Infusions
Groups:
- SCIG Treatment: IgPro20 was administered subcutaneously with the first SC IgPro20 infusion starting 1 week after the last IVIG dose. Subjects were treated with weekly SC IgPro20 infusions for a 12-week wash-in/wash-out period followed by a 12-week efficacy period. The IgPro20 dose was to be equal to the weekly equivalent dose of the previous IVIG IgG treatment.
Arm/Group | IVIG Treatment | SCIG Treatment
Number analyzed (Participants) | 25 | 25
Number analyzed (Infusions) | 75 | 584
AEs per infusion
  All AEs | 0.653 | 0.457
  At Least Possibly Related AEs | 0.027 | 0.296
  Serious AEs | 0 | 0.002
  At Least Possibly Related and Serious AEs | 0 | 0

11. Secondary Outcome: Rate of Mild, Moderate, or Severe Local Reactions
Description: In addition to the standard MedDRA System Organ Class (SOC) AE assignments, the category of 'local reactions' was defined to provide the possibility for a combined analysis of local reactions and included AEs of: infusion site discomfort, infusion site erythema, infusion site haemorrhage, infusion site induration, infusion site inflammation, infusion site pain, infusion site pruritus, infusion site swelling, injection site erythema, injection site extravasation, injection site induration, injection site irritation, injection site pain, injection site pruritus, injection site swelling, and puncture site reaction.
  Mild AE: Symptoms are easily tolerated and there is no interference with daily activities; Moderate AE: Discomfort enough to cause some interference with daily activities; Severe AE: Incapacitating with inability to work or do usual activity.
Time Frame: For the duration of the study, up to 36 weeks
Population: The SDS comprised all subjects treated with the study drug.
Measure: Number; unit: AEs per infusion
Units Other Than Participants: Infusions
Arm/Group | IVIG Treatment | SCIG Treatment
Number analyzed (Participants) | 25 | 25
Number analyzed (Infusions) | 75 | 584
AEs per infusion
  Mild Local Reactions | 0 | 0.274
  Moderate Local Reactions | 0 | 0
  Severe Local Reactions | 0 | 0

ADVERSE EVENTS:
Time Frame: For the duration of the study, up to 36 weeks
Description: The safety data set comprised all subjects treated with the study drug. All SAEs are presented including a pre-treatment SAE of gastroenteritis. In Other AEs, non-serious AEs starting at or after the first study drug infusion are presented. A total of 75 IVIG and 584 SCIG infusions of IgPro20 were administered to 25 subjects during the study.
Groups:
- IVIG Treatment: Study subjects were treated with their IVIG therapy with 3- or 4-weekly schedules for 3 dosing cycles (9 to 12 weeks; before being switched to SCIG treatment with IgPro20).
Arm/Group | IVIG Treatment | SCIG Treatment
Serious Adverse Events (participants affected / at risk) | 1/25 | 1/25
Other Adverse Events (participants affected / at risk) | 20/25 | 24/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IVIG Treatment (N=25) | SCIG Treatment (N=25)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) — This SAE occurred between screening and the first IVIG dose and was thus non-treatment-emergent.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IVIG Treatment (N=25) | SCIG Treatment (N=25)
Dental caries (Gastrointestinal disorders) | 1 (1) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Local reactions (General disorders) | 0 (0) | 20 (160) — Local reactions cover MedDRA PTs: infusion site: discomfort, erythema, haemorrhage, induration, inflammation, pain, pruritus, swelling; injection site: erythema, extravasation, induration, irritation, pain, pruritus, swelling; puncture site reaction.
Bronchitis (Infections and infestations) | 0 (0) | 3 (3)
Conjunctivitis infective (Infections and infestations) | 1 (1) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 3 (5)
Influenza (Infections and infestations) | 4 (4) | 4 (4)
Nasopharyngitis (Infections and infestations) | 5 (8) | 11 (21)
Sinusitis (Infections and infestations) | 0 (0) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 5 (8)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 3 (7)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 3 (3) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (9)
Malaise (General disorders) | 2 (2) | 1 (2)
Pharyngitis (Infections and infestations) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
CSL agreements and restrictions on publishing may vary with individual investigators; however, CSL will not prohibit any investigator from publishing. CSL supports the publication of results from all centers of a multi-center trial and generally requires that reports based on single-site data not precede the primary publication of the entire clinical trial.